CLINICAL TRIAL: NCT02730962
Title: Interventional Bioremediation of Microbiota in Metabolic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Delays in IND approval caused a lack of funding to conduct the trial.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GI-2015-22791
Record Dates: First submitted 2016-03-16; First posted 2016-04-07 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Pre-Diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Vancomycin; Neomycin; Clindamycin; Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotics prior to FMT (Experimental): One week prior to FMT, a course of three oral antibiotics are taken: Vancomycin 500mg, Neomycin 1000mg, and Clindamycin 300mg.
  Interventions: Drug: Vancomycin; Drug: Neomycin; Drug: Clindamycin; Procedure: Fecal Microbiota Transplantation
- Placebo prior to FMT (Placebo Comparator): One week prior to FMT, a course of three sugar pills identical to each antibiotic.
  Interventions: Other: Placebo; Procedure: Fecal Microbiota Transplantation

INTERVENTIONS:
Drug: Vancomycin — Vancomycin 3 times a day for 7 days
  Arms: Antibiotics prior to FMT
Other: Placebo — Placebo pills identical in appearance to each antibiotics to be taken on the same schedule as each antibiotic
  Arms: Placebo prior to FMT
Drug: Neomycin — Neomycin 3 times a day for 1 day
  Arms: Antibiotics prior to FMT
Drug: Clindamycin — Clindamycin 3 times a day for 5 days
  Arms: Antibiotics prior to FMT
Procedure: Fecal Microbiota Transplantation — FMT conducted via colonoscopy

SUMMARY:
The purpose of this study is to determine whether changing the microbial composition in the colon can improve metabolism of sugar in people who are on the verge of developing diabetes (pre-diabetics). Study participants will undergo a fecal microbiota transplantation (FMT) using material from lean donors, as well as a series of tests prior to and after the transplant. The investigators will examine any changes in fecal bacterial composition associated with FMT and determine if any observed changes have an influence on blood sugar metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent
2. Ambulatory and community dwelling
3. Age 18 - 70 years of age
4. Able and willing to comply with the study schedule and procedures
5. Pre-diabetic with fasting blood glucose > 100 mg/dL and/or blood glucose 140-200 mg/dL 2-hours after ingestion of 75 gm glucose and/or Hemoglobin A1c > 5.7-6.5 percent

Exclusion Criteria:

1. Serious, concomitant illness that, in the opinion of the Investigator, would interfere with evaluation of safety or efficacy, or put the subject at risk of harm from study participation.
2. Known inflammatory bowel disease (Crohn's disease, ulcerative colitis, lymphocytic colitis).
3. Current abnormal liver tests that may be attributed to a cause other than non-alcoholic liver disease. Note: These exclusionary conditions may include viral hepatitis, alcoholic liver disease, hemochromatosis, Wilson's disease, medication-induced liver test abnormalities, celiac disease.
4. Renal insufficiency, defined as creatinine ≤ 1.25 mg/dL
5. Significant alcohol use, defined as > 20 g/day in females and > 30 g/day in males for a period of 3 months within one year prior to screening.
6. Underlying chronic gastrointestinal disease that can cause diarrhea, including short bowel syndrome, diarrhea-predominant irritable bowel syndrome, malabsorption, celiac disease.
7. History of partial or complete colectomy.
8. History of malabsorptive bariatric surgery.
9. Use of insulin or hypoglycemic medications.
10. History of anaphylactic food allergies, e.g., peanuts, seafood.
11. Food intolerances and allergies, including gluten sensitivity, lactose intolerance, and intolerance of high fiber dietary content.
12. Symptomatic problems associated with intestinal gas and bloating.
13. Irritable bowel syndrome, including diarrhea-dominant, constipation-dominant, and mixed.
14. Functional GI disorder.
15. Unable to tolerate a colonoscopy.
16. Presence of an indwelling intravenous line.
17. Infection requiring antibiotics other than the conditioning antibiotics during the study period.
18. Inability to take vancomycin, neomycin, and clindamycin antibiotics prior to FMT due to known hypersensitivity or intolerance.
19. Major genetic immune dysfunction (e.g., common variable immune deficiency).
20. Acquired immune deficiencies due to infections such as HIV.
21. Immunosuppressive medications including one of the following: systemic corticosteroids, calcineurin inhibitors, thiopurines, methotrexate, biologics (e.g., anti-tumor necrosis factor drugs), cancer chemotherapy.
22. Planned use of oral probiotics while on study.
23. Planned or ongoing chemotherapy for malignancy.
24. Planned antibiotic therapy within the period of the study, e.g., perioperative antibiotics.
25. Pregnant or lactating. Female participants of child-bearing age and their partners will be counseled on contraceptive measures to prevent pregnancy during the study period.
26. History of drug or alcohol abuse in the past 2 years.
27. Currently participating in another clinical study.
28. Legally incompetent and unable to understand the study's purpose, significance and consequences, and to make decisions accordingly.
29. Presence of metal implants, such as surgical clips or pacemakers, which will preclude performance of MRI tests.
30. Inability to undergo MRI testing for any reason, e.g., claustrophobia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Khoruts, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antibiotics Prior to FMT | Placebo Prior to FMT
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibiotics Prior to FMT | Placebo Prior to FMT | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (9.63) | 46.6 (7.95) | 44.9 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Insulin sensitivity measured by standard euglycemic insulin clamp.
Time Frame: 10 weeks
Population: Due to errors in formulation of the euglycemic insulin clamp solutions, insulin sensitivity data is not able to be analyzed.
Arm/Group | Antibiotics Prior to FMT | Placebo Prior to FMT
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Microbiome Composition
Description: Outcome is reported as the Shannon alpha diversity index (unitless measure) at baseline and 7 days post FMT.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: unitless measure
Arm/Group | Antibiotics Prior to FMT | Placebo Prior to FMT
Number analyzed (Participants) | 7 | 5
unitless measure
  Baseline | 3.3 (0.5) | 3.3 (0.5)
  7 days post FMT | 3.3 (0.5) | 1.2 (0.2)

3. Secondary Outcome: Changes in Fecal Bacterial Composition Associated With FMT Overall Antibiotic and Placebo Conditioning Groups) by Laboratory Analysis.
Description: Microbiome composition was assessed post FMT using fecal DNA extraction and sequences. Outcome is reported as the change in relative abundance of the family Ruminococcaceae.
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: percent relative abundance
Arm/Group | Antibiotics Prior to FMT | Placebo Prior to FMT
Number analyzed (Participants) | 7 | 5
percent relative abundance | 5 (2) | 17 (1)

4. Secondary Outcome: Adverse Event Rates
Description: Outcome is reported as a patient self report of adverse events over 10 weeks.
Time Frame: 10 weeks
Measure: Number; unit: Number of adverse events
Arm/Group | Antibiotics Prior to FMT | Placebo Prior to FMT
Number analyzed (Participants) | 7 | 5
Number of adverse events | 6 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected at each study visit during study participation, which was approximately 3-4 months, and collected again at a 6 month follow up visit after study completion.
Arm/Group | Antibiotics Prior to FMT | Placebo Prior to FMT
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/5
Other Adverse Events (participants affected / at risk) | 6/7 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antibiotics Prior to FMT (N=7) | Placebo Prior to FMT (N=5)
Clostridium Difficile Infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antibiotics Prior to FMT (N=7) | Placebo Prior to FMT (N=5)
Diarrhea (Gastrointestinal disorders) | 5 (9) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (1)
Fatigue (General disorders) | 4 (4) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Superficial Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT02730962/Prot_SAP_000.pdf